CLINICAL TRIAL: NCT03731884
Title: Proteomic and Lipidomic Profiling of Coronary Thrombus in Acute Myocardial Infarction
Brief Title: Proteomic Profiling of Coronary Thrombus in Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G. d'Annunzio University (Other)
Collaborators: Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Marco Zimarino, Principal investigator, G. d'Annunzio University
Other Study IDs: PROTEOTHR18
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Acute Myocardial Infarction; STEMI - ST Elevation Myocardial Infarction
Keywords: Coronary thrombus; Proteomics; Lipidomics; Thrombus aspiration
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lyophilized thrombus extracted by thrombus-aspiration in patients with acute myocardial infarction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elapsed time of onset-of-pain-to-PCI <3 hours: Patients with AMI undergoing percutaneous coronary intervention (PCI) prior to 3 hours from the onset of symptoms
  Interventions: Other: Time from the onset of symptoms to PCI
- Elapsed time of onset-of-pain-to-PCI >3 hours: Patients with AMI undergoing percutaneous coronary intervention (PCI) after at least 3 hours from the onset of symptoms
  Interventions: Other: Time from the onset of symptoms to PCI

INTERVENTIONS:
Other: Time from the onset of symptoms to PCI — Patients will be divided in two groups according to the time from the onset of symptoms to PCI

SUMMARY:
ST-elevation myocardial infarction (STEMI) is mostly caused by the rupture or the erosion of a vulnerable atherosclerotic plaque, initiating with intraluminal thrombosis and resulting in total occlusion of the coronary artery. Thrombus formation is a complex and dynamic process involving flow, blood cells and several plasma proteins, and it has not been clearly elucidated. To define - through proteomic approach - the composition of occluding thrombus and its time changes in patients with STEMI, trying to identify novel biomarkers of coronary thrombosis.

DETAILED DESCRIPTION:
Ischemic heart disease is the leading contributor to the worldwide burden of disease, as assessed on the basis of disability-adjusted life-years.

ST-Elevation Myocardial Infarction (STEMI) is associated with a coronary occlusive thrombosis in 90% of patients, non-ST Elevation Myocardial Infarction (NSTEMI) only in 26% of cases. In this regard, increasing attention is given to the composition of coronary thrombus. In acute STEMI, platelet and fibrin content in the occlusive thrombus is highly dependent on ischemia time, thus one can infer that this may have a substantial impact on the efficacy of drugs or devices used for coronary reperfusion.

Among several circulating cell types - platelets, erythrocytes, monocytes, and neutrophils - as well as plasma molecules, modulating the thrombosis process, platelets constitute the major cellular component of the thrombus and their activation is essential for thrombus formation. Although the role of platelets in thrombosis has been deeply characterized, the molecular mechanisms underlying platelet activation and focal adhesion within human coronary thrombi, the composition, time changes of the occluding thrombus and its interaction with the other cells have not been clearly elucidated, mainly due to the difficult accessibility to the thrombotic material. Thrombus aspiration, although having a controversial role as an adjunctive strategy in primary percutaneous coronary intervention (PCI) for STEMI and NSTEMI, relies on the extraction of occlusive thrombi by an aspiration catheter, advanced in the coronary arterial tree and constitutes a unique opportunity for obtaining coronary thrombi from patients suffering from AMI.

Defining variable molecular pathways responsible for thrombus formation according to time lapse and pathophysiology may pave the way to newer therapeutic strategies.

Hypothesis of the study Coronary thrombus undergoes significant modification according to the pathophysiology of formation (erosion, plaque rupture or metal strut exposure) and time-lapse from symptom onset.

The exact definition the molecular composition of coronary thrombus and of its proteomic and metabolomics patterns may identify the target of newer therapeutic strategies.

Aims of the study are: to elucidate the molecular composition of coronary thrombus in AMI, to understand, at molecular level, phenotypic alteration related to thrombus formation, to highlight new potential factors involved in disease's onset or related to time of thrombus formation.

A consecutive series of patients admitted for an ACS, with either STEMI and occluded infarct-related artery or NSTEMI and visible thrombus in the culprit artery will be deemed suitable for thrombus aspiration. PCI will be performed with a standard procedure, with either femoral or radial access. All patients will be receiving acetylsalicylic acid (100 mg daily) and a P2Y12 inhibitor - clopidogrel (600 mg, then 75 mg daily), prasugrel (60 mg, then 10 mg daily) or ticagrelor (180 mg daily). After insertion of the arterial sheath, every patient will receive 70 IU/kg of heparin.

After guidewire positioning across the lesion, the thrombus aspiration system will be advanced with gentle suction and several passages will be performed through the culprit lesion.

The lyophilized thrombus from each patient enrolled will undergo to extensive molecular characterization in term of proteins, metabolites (Amino Acids and Acylcarnitines) and polar lipids.

Polar metabolites and lipids from thrombus will be extracted and analyzed following a validated methodology: 5 mg of wet thrombus will be added to a 330 μL of methanol solution containing deuterated internal standards of amino acids and carnitines and lyso-sphingomyelin 100 µg/ml as internal standard for lipidomics. These solutions will be incubated at 45 °C for 50 min and finally divided into two aliquots. The first one will be used to analyze amino acids and acyl-carnitines following our LC-MS/MS method already used in the analysis of CSF as previously reported. The second aliquot will be employed to screen phospholipids by LC-MS/MS. Data obtained will be quantified using MarkerLynx and NeoLynx software, and statistically investigated using GraphPad Prism, Simca P+ and MetaboAnalyst software.

The lyophilized thrombus will be digested by Filter Aided Sample Prep (FASP) protocol. Then, instrumental triplicates will be acquired for each sample by a platform nanoLC-ESI-QTOF-MS/MS performing label free shotgun proteomics experiments in order to identify, and simultaneously, quantify expressed proteins as already reported. The result of this study will be a list of expressed proteins during coronary thrombus in acute myocardial infarction, that may be used for bioinformatics analysis.

Data will be processed by a dedicated software (Profile Analysis, Bruker, Markerlynx). Highlighted metabolites/proteins will be identified by database and by fragmentation analysis.

Specifically for metabolomics and lipidomics, the data will be processed to obtain peak deconvolution and alignment, denoise and Total Ion Count normalization to give a table of mass pairs with associated relative intensities for all the detected peak for each sample analyzed. Then, the data matrix will be used for multivariate Analysis (PCA; PLS-DA) using SIMCA-P + 11.0 (Umetrics AB, Umeå, Sweden).

By multi-omics researches and data processing, it will be available a panel of interesting molecules as a framework for each clinical group studied. These biological compounds will be then subjected to an in-silico analysis to rebuild their functional implications in the physiology and molecular homeostasis of coronary thrombus in acute myocardial infarction. To perform such a meta-analysis of the data we will mainly use Ingenuity Pathways Analysis (IPA), (Ingenuity Systems, Mountain View, CA). Through the Pathways analysis and the Gene Ontology it will be possible to identify the metabolic pathways and the secondary genes/proteins inhibited and/or stimulated for a specific phenotype and consequently classify potential effectors molecules and/or pharmacological target.

ELIGIBILITY:
Inclusion Criteria:

* patients with STEMI and occluded infarct-related artery or NSTEMI and visible thrombus deemed suitable for thrombus aspiration

Exclusion Criteria:

* thrombus aspiration not performed or unsuccessfull

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients admitted for an ACS, with either STEMI and occluded infarct-related artery or NSTEMI and visible thrombus in the culprit artery will be deemed suitable for thrombus aspiration. PCI will be performed with a standard procedure, with either femoral or radial access.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change through time in thrombus proteomic composition | within 24 hours
  Compare concentrations of different protein types in the supernatant of thrombus from patients with STEMI<3hs vs <3hs, through proteomic approaches

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zimarino, MD, PhD, Principal Investigator — G. D'Annunzio University. Institute of Cardiology; Damiana Pieragostino, Study Chair — Department of Medical, Oral and Biotechnological Sciences, G. d'Annunzio University - Chieti
Locations (1):
- Santissima Annunziata Hospital, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pieragostino D, D'Alessandro M, di Ioia M, Rossi C, Zucchelli M, Urbani A, Di Ilio C, Lugaresi A, Sacchetta P, Del Boccio P. An integrated metabolomics approach for the research of new cerebrospinal fluid biomarkers of multiple sclerosis. Mol Biosyst. 2015 Jun;11(6):1563-72. doi: 10.1039/c4mb00700j. PMID 25690641
- [Background] Del Boccio P, Pieragostino D, Di Ioia M, Petrucci F, Lugaresi A, De Luca G, Gambi D, Onofrj M, Di Ilio C, Sacchetta P, Urbani A. Lipidomic investigations for the characterization of circulating serum lipids in multiple sclerosis. J Proteomics. 2011 Nov 18;74(12):2826-36. doi: 10.1016/j.jprot.2011.06.023. Epub 2011 Jul 4. PMID 21757039
- [Background] Zimarino M, Angeramo F, Prasad A, Ruggieri B, Malatesta S, Prati F, Buttitta F, De Caterina R. Reduction of atherothrombotic burden before stent deployment in non-ST elevation acute coronary syndromes: Reduction of myocardial necrosis achieved with nose-dive manual thrombus aspiration (REMNANT) trial. A volumetric intravascular ultrasound study. Catheter Cardiovasc Interv. 2016 Nov;88(5):716-725. doi: 10.1002/ccd.26301. Epub 2015 Nov 3. PMID 26527239